CLINICAL TRIAL: NCT02887768
Title: Cardiac Infarct Repair Using CorMatrix®-ECM: Clinical Feasibility Study
Brief Title: Epicardial Infarct Repair Using CorMatrix®-ECM: Clinical Feasibility Study
Acronym: EIR
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Corvivo Cardiovascular, Inc. (Industry)
Responsible Party: Principal Investigator, Dr. Paul Fedak, Professor and Cardiac Surgeon, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB14-1715
Record Dates: First submitted 2016-04-02; First posted 2016-09-02 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Acute Coronary Syndrome; Heart Failure
MeSH Terms: conditions — Acute Coronary Syndrome; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Epicardial Infarct Repair with CorMatrix-ECM in addition to coronary artery bypass grafting
  Interventions: Device: Epicardial Infarct Repair with CorMatrix-ECM; Procedure: Coronary Artery Bypass Grafting Surgery

INTERVENTIONS:
Device: Epicardial Infarct Repair with CorMatrix-ECM — CorMatrix-ECM-biomaterial will be surgically applied to the epicardial surface of the infarct myocardium at the time of coronary artery bypass surgery
  Other Names: SIS-ECM (small intestine submucosa extracellular matrix)
Procedure: Coronary Artery Bypass Grafting Surgery — All participants will undergo standard coronary artery bypass grafting surgery to treat coronary artery disease
  Other Names: Aorto-coronary bypass surgery

SUMMARY:
Epicardial Infarct Repair with CorMatrix-Extracellular Matrix (ECM) is an open-label, non-randomized, feasibility pilot study. Following ischemic injury the ECM of the heart adversely remodels leading to cardiac fibrosis, left ventricular (LV) dilatation and subsequent heart failure. Preclinical evidence demonstrates that epicardial infarct repair with CorMatrix-ECM restores the damaged ECM, prevents LV dilatation and improves myocardial performance. This study will interrogate epicardial infarct repair in patients undergoing coronary artery bypass grafting (CABG) surgery within 6 weeks following acute myocardial infarction as an adjunct to surgical revascularization. Patients will be evaluated for markers of cardiac function and left ventricular remodelling using cardiac magnetic resonance imaging (MRI). Adverse events will be monitored to ensure safety.

DETAILED DESCRIPTION:
RATIONALE: Following ischemic injury the extracellular matrix (ECM) of the heart adversely remodels leading to cardiac fibrosis, left ventricular (LV) dilatation and subsequent heart failure. Preclinical evidence suggests that the epicardial application of a healthy biologic ECM may reverse the adverse ECM remodeling that takes place following ischemic injury preventing LV dilatation and subsequent heart failure. The investigators have demonstrated that epicardial infarct repair with CorMatrix-ECM restores the damaged ECM, prevents LV dilatation and improves myocardial performance. The investigators believe that epicardial infarct repair may not only restrain the infarcted myocardium to prevent infarct expansion and LV dilatation, but owing to it's biologic nature, help to provide a healthy ECM environment restoring ECM homeostasis and architecture. The investigators therefore propose clinical investigation epicardial infarct repair in patients undergoing coronary artery bypass grafting (CABG) surgery within 6 weeks following acute myocardial infarction as an adjunct to surgical revascularization. This is a patient population commonly referred for CABG surgery. While complete surgical revascularization can prevent further ischemic insult and salvage stunned or hibernating myocardium, it does not restore function to the infarcted myocardium resulting from the acute ischemic injury. The investigator's previous studies suggest that epicardial infarct repair as an adjunct to CABG surgery in this patient population may help improve myocardial function in this previously untreatable territory.

STUDY DESIGN: This is an open-label, non-randomized, feasibility pilot study

PRIMARY OBJECTIVE:

• To evaluate the feasibility of epicardial infarct repair performed with CorMatrix-ECM as an adjunct to CABG surgery in patients undergoing surgery during the subacute period following myocardial infarction (MI).

SECONDARY OBJECTIVES:

* To evaluate the feasibility of identifying the infarct area to be treated by epicardial infarct repair and measure regional function and tissue characteristics within the treated area using cardiac magnetic resonance (CMR) imaging.
* To evaluate the safety of epicardial infarct repair performed with CorMatrix-ECM as an adjunct to CABG surgery.

NUMBER OF SUBJECTS: Eight

TEST PRODUCT, DOSE, AND ROUTE OF ADMINISTRATION: CorMatrix-ECM will be surgically applied to the epicardial surface of the anterior LV wall at the time of coronary artery bypass surgery.

CONTROL PRODUCT, DOSE AND ROUTE OF ADMINISTRATION: No control group will be performed in this pilot trial.

DURATION OF SUBJECT PARTICIPATION AND DURATION OF STUDY: Subjects will be involved in the study for up to 6 months.

Screening/Enrollment: 0-6 weeks between acute coronary syndrome presentation and CABG surgery.

Treatment: Day of CABG surgery. Follow-up: 6 months postoperatively. Total duration of the study is expected to be 9 months. Three months for subject enrollment and 6 months for final subject follow-up.

CONCOMMITANT MEDICATIONS:

Prohibited: Immunosuppressive medications (including steroids). Allowed: Any other medications.

FEASIBILITY EVALUATIONS: Feasibility will be accessed through qualitative evaluation by the performing surgeon and successful measurement of cardiac function and tissue characterization by CMR.

PRIMARY ENDPOINT:

• Feasibility of epicardial infarct repair performed with CorMatrix-ECM as an adjunct to CABG surgery in patients undergoing surgery during the subacute period following myocardial infarction (MI) evaluated by the performing surgeon though qualitative observation.

SECONDARY ENDPOINTS:

* Feasibility of measuring regional myocardial function and tissue characteristics within the treated area using cardiac magnetic resonance (CMR) imaging.
* The safety of epicardial infarct repair performed with CorMatrix-ECM.

SAFETY EVALUATIONS :

Adverse events including: all cause mortality; cardiovascular mortality; MACCE; major bleeding events; primary surgical site infection; and myocardial constriction will be recorded.

RATIONALE FOR NUMBER OF STUDY SUBJECTS: This is a pilot study designed to access the feasibility of performing epicardial infarct repair with CorMatrix-ECM in subacute MI patients going for CABG surgery, the feasibility of measuring cardiac function and various tissue characteristics within the treated myocardium by CMR in this patient population, and the safety of epicardial infarct repair performed at the time of CABG surgery. Given the preliminary nature of this study 8 subjects will be tested to confirm feasibility and inform future randomized control trial study design.

ELIGIBILITY:
Inclusion Criteria:

* The patient has been diagnosed with an acute STEMI or NSTEMI (confirmed by ST changes on serial ECG, elevated troponin, coronary artery stenosis or occlusion identified by angiography, and a wall motion abnormality identified by angiography or echocardiography)
* The patient is scheduled to undergo coronary artery bypass surgery within 6 weeks of the acute event.
* The patient does not possess any contraindication for CMR.
* The patient is greater then 35-years of age, English speaking, and capable of giving informed consent.
* The patient is geographically accessible and willing to return for all follow-up investigations and clinical visits associated with study.

Exclusion Criteria:

* The patient is over the age of 75 years.
* The patient has previous MI (other than the qualifying event) and/or has scar or non-viable myocardium identified by CMR in any other LV territory.
* The patient is undergoing other cardiac surgery (i.e. concurrent cardiac valve, or aortic surgery).
* The patient requires emergency surgery (i.e. operative intervention (CABG or ventricular assist device) within 24-hrs of assessment).
* The patient has undergone previous cardiac surgery.
* The patient's postsurgical life expectancy is less than 45 days, in the investigator's opinion.
* The patient is of excessively poor baseline health, health-related quality of life, or physical functioning that would preclude a reasonable expected post-operative recovery.
* The patient has received radiotherapy to the chest wall, is receiving immunosuppressive therapy, or is in any way immunocompromised.
* The patient has a history of malignancy within the past year (other than squamous or basal cell carcinoma, which has been treated without evidence of recurrence).
* The patient has a recent history of drug or alcohol abuse.
* The patient has within 30-days of enrollment or is at anytime during this study participating in any other drug or device study.
* The patient has a known allergy to the CorMatrix-ECM material or any component of the material.
* Absence of non-viable myocardium within the LV on CMR.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-01; Primary Completion 2017-07 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
The number of patients in which the study intervention is successfully completed | 6 weeks
  Feasibility will be accessed through qualitative evaluation by the performing surgeon. Successful application of CorMatrix-ECM to the infarcted myocardium at the time of coronary artery bypass grafting surgery will be deemed as successful completion of the study intervention.

SECONDARY OUTCOMES:
The number of patients in which the target myocardium can be successfully identified at the time of surgery | 6 weeks
  The infarct area will be identified by CMR using a standard late gadolinium enhancement protocol and the feasibility of correlating the CMR images with the surgical anatomy will be qualitatively evaluated by the performing surgeon.
The number of patients in which regional myocardial function and tissue characteristics are successfully measured by CMR | 6 months
  The feasibility of evaluating both regional function and tissue characteristics will be confirmed by successful measurement of left ventricular volume, ejection fraction, regional wall motion, myocardial edema, myocardial fibrosis, myocardial tissue viability and myocardial strain using cardiac magnetic resonance (CMR).
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul WM Fedak, MD, PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data will only be shared with that patient. De-identified and compiled data will be used for analysis and publication.

REFERENCES:
- [Result] Mewhort HE, Turnbull JD, Satriano A, Chow K, Flewitt JA, Andrei AC, Guzzardi DG, Svystonyuk DA, White JA, Fedak PW. Epicardial infarct repair with bioinductive extracellular matrix promotes vasculogenesis and myocardial recovery. J Heart Lung Transplant. 2016 May;35(5):661-70. doi: 10.1016/j.healun.2016.01.012. Epub 2016 Jan 15. PMID 26987597
- [Result] Mewhort HE, Turnbull JD, Meijndert HC, Ngu JM, Fedak PW. Epicardial infarct repair with basic fibroblast growth factor-enhanced CorMatrix-ECM biomaterial attenuates postischemic cardiac remodeling. J Thorac Cardiovasc Surg. 2014 May;147(5):1650-9. doi: 10.1016/j.jtcvs.2013.08.005. Epub 2013 Sep 26. PMID 24075463
- See also: Article: Epicardial infarct repair with bioinductive extracellular matrix promotes vasculogenesis and myocardial recovery — http://www.jhltonline.org/article/S1053-2498(16)00059-0/fulltext